CLINICAL TRIAL: NCT00580034
Title: Allogeneic (Allo) Non-Myeloablative Stem Cell Transplantation (SCT) Utilizing Mis-Matched Family Member Stem Cells Purged Using Campath-1H
Brief Title: Allo Non-Myeloablative SCT Utilizing Mis-Matched Family Member Stem Cells Purged Using Campath
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: David Rizzieri, MD (Other)
Collaborators: Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Sponsor-Investigator, David Rizzieri, MD, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00009528
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Lymphoma; Myeloma; Leukemia; Myelodysplasia; Solid Tumors
Keywords: Allogeneic Stem Cell Transplantation, Campath, HLA-Matched
MeSH Terms: conditions — Lymphoma; Neoplasms, Plasma Cell; Leukemia; Anemia, Refractory, with Excess of Blasts

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Campath Purged Non-myeloablative ASCT (Experimental): Campath Purged Non-myeloablative Allo Stem Cell Transplant (ASCT) in lymphoma, myeloma, or marrow failure: leukemia or myelodysplasia; and solid tumors
  Interventions: Drug: Campath Purged Non-myeloablative ASCT
- Donor Apheresis (Other): Donor must be a sibling, half sibling, parent, child or first cousin familial relationship and 3-5/6 Human Leukocyte Antigen matched related to subject. They must not have any medical condition which would make apheresis and G-CSF administration more than a minimal risk, and should have the following:
  1. Adequate cardiac function by history and physical examination
  2. bilirubin and hepatic transaminases < 2.5 x upper limit of normal
  3. normal hematologic parameters Females should have a negative serum pregnancy test.
  Interventions: Procedure: Donor Apheresis

INTERVENTIONS:
Drug: Campath Purged Non-myeloablative ASCT — Preparative regimen: Begins on day -5 and consist of 4 days of daily fludarabine at 30 mg/m2/d infused over 30 minutes, cyclophosphamide 500 mg/m2/d infused over 1 hour, 5 days of Campath-1H at 20 mg/d in 250 ml of D5 normal saline or normal saline infused over 3 hours.
  Patient Evaluation: Will occur 2-3 times per week by physical exam for toxicity through day 45.
  Arms: Campath Purged Non-myeloablative ASCT
Procedure: Donor Apheresis — Donor will receive Granulocyte colony-stimulating factor (G-CSF) 10-16 mcg/kg/d subcutaneously (dose will be rounded to the nearest whole vial size and may be divided into twice daily dosing). Granulocyte-macrophage colony-stimulating factor (GM-CSF) 15 mcg/kg/d subcutaneous or similar growth factor for donor mobilization. Donors will receive at least 3-6 doses of daily growth factor until adequate cells are mobilized.
  Arms: Donor Apheresis

SUMMARY:
Allogeneic transplantation is used to treat many malignant and non-malignant diseases, though the potential toxicities of the procedure remain high. We and others have shown that a less toxic preparative regimen allows reliable allogeneic engraftment for allogeneic transplantation.

The primary purpose of this treatment trial is to follow patients undergoing allogeneic transplantation for long term outcomes. The regimen used has been tested in our prior phase I / II trial which has completed accrual. The issues of engraftment and rate of graft versus host disease have been answered and our success has led to this regimen being a standard approach for less toxic allogeneic therapy.

DETAILED DESCRIPTION:
Allogeneic bone marrow transplantation may cure or ameliorate illnesses of many types; however the toxicity of the procedure limits its broad applicability. Hematologic malignancies of all types have shown responses. Those with marrow failure, such as aplasia, and hemoglobinopathies have further shown responses in multiple trials as well. Even patients with certain solid tumors, such as breast, renal cell, and melanoma have shown partial or complete responses to allogeneic therapy. The limiting effect of the historical methods of aggressive induction for allogeneic therapy were extremely toxic, requiring limiting those offered allogeneic therapy to the healthiest of the ill patients. Work over the last decade has shown that less toxic agents targeting the immune system effectively allowed engraftment with less effects on the patient's liver, lungs, and other vital organs. We and others have completed multiple trials showing the effective use of these less toxic, non-myeloablative, regimens for allogeneic therapy. Trials with fludarabine and cyclophosphamide at standard doses (patients are not ablated and recover blood counts in 2 weeks) allow for 80% of patients to engraft donor cells. Some groups have added low doses of radiation to this combination, with 80-100% allogeneic engraftment. The lessened toxicity of this approach has been confirmed in multiple studies, including our own data with the specific schema in this treatment plan reviewed below. Phase I results with this combination: Our group has combined the above combination of fludarabine and cyclophosphamide with the antibody CAMPATH 1H. This antibody is given to the patient to purge the immune system and prevent rejection. It also purges the T cells in the donated stem cells to minimize graft versus host disease (GVHD). This approach has been proven successful in multiple trials using standard more toxic ablative procedures. Our approach over the last 3 years has been very successful using this antibody with the less toxic non-myeloablative procedure and our trials have completed.

The primary purpose of this treatment trial is to follow patients undergoing allogeneic transplantation for long term outcomes. The regimen used has been tested in our prior phase I / II trial which has completed accrual. The issues of engraftment and rate of graft versus host disease have been answered and our success has led to this regimen being a standard approach for less toxic allogeneic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have their pathology reviewed and the diagnosis confirmed.
* Performance status (PS) must be Cancer and Leukemia Group B (CALGB) PS 0, 1, or 2
* Patients must have a 3-5/6 Human leukocyte antigen (HLA)-matched related donor who is evaluated and deemed able to provide peripheral blood progenitor cells (PBPCs) and/or marrow by the transplant team.
* HIV antibody negative.
* Patients must test negative for serum beta-human chorionic gonadotropin (hCG) and must agree to use some form of adequate birth control during the periods they receive chemotherapy and any post-chemotherapy medications related to the transplant.
* Patients must be 17 years of age or greater.
* Patients must also have a resting Multi Gated Acquisition Scan (MUGA) and/or echocardiography (ECHO) and pulmonary function tests (PFTs) with testing of diffusing capacity of the lung for carbon monoxide (DLCO) performed before transplant and found to be acceptable according to the treating institution's guidelines. The required minimum standards include MUGA and/or ECHO showing an ejection fraction (EF) of 40% and PFTs showing DLCO of 40%. Those with an EF 40-50%, undergo cardiac evaluation and consultation. Also, those with DLCO 40-50%, undergo pulmonary evaluation and consultation.
* Specific populations for each disease category:

  * Hematologic malignancies Those with high risk or relapsed hematologic malignancy (including myeloid and lymphoid leukemias and lymphomas, myeloma or myelomatous like diseases, myeloproliferative disease, myelodysplasia). Those with good risk disease (first remission acute myeloid leukemia (AML) with myelomonocytic together with bone marrow eosinophilia (M4eos) - inversions in chromosome 16, promyelocytic (M3) AML with translocations in chromosomes (15;17); or translocations in chromosomes (8;21) in first remission are not eligible).
  * Bone marrow failure:

    * Those specifically with idiopathic or secondary moderate, severe or very severe aplastic anemia (idiopathic or secondary) according to the accepted 'Camitta criteria' would be candidates.
    * Those with diseases known to lead to severe marrow failure are eligible as well. These include those with myelofibrosis or Paroxysmal nocturnal hemoglobinuria (PNH).
  * Solid Tumors:

    * Patients must have had a biopsy confirming disease recurrence (metastases) at some point in their history, unless the patient presented with metastatic disease, in which case the initial primary site biopsy is adequate.
* Patients with renal cell cancer, or melanoma will be eligible for this approach at this time. Patients will have had documented metastatic disease at some time in the past. Patients who are in remission or with residual disease after prior therapy for their metastatic disease are eligible, as there is no accepted cure for these patients with metastatic disease.
* Breast Cancer- Patients will have had documented metastatic disease at some time in the past. Patients who are in remission or with residual disease after prior therapy for their metastatic disease are eligible. Patient must have failed at least one chemotherapy regimen for their metastatic disease and 1 hormonal agent if they are receptor positive.

Exclusion Criteria:

* Pregnant or lactating women,
* Patients with other major medical or psychiatric illnesses which the treating physician feels could seriously compromise tolerance to this protocol, and
* Leukemia patients in first remission with good risk cytogenetics for leukemia [t(15;17); t(8,22)]

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2003-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Rizzieri, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Health Systems, Durham, North Carolina, United States

REFERENCES:
- [Result] Rizzieri DA, Dev P, Long GD, Gasparetto C, Sullivan KM, Horwitz M, Chute J, Chao NJ. Response and toxicity of donor lymphocyte infusions following T-cell depleted non-myeloablative allogeneic hematopoietic SCT from 3-6/6 HLA matched donors. Bone Marrow Transplant. 2009 Feb;43(4):327-33. doi: 10.1038/bmt.2008.321. Epub 2008 Oct 13. PMID 18850014

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in February, 2003 and ended in February, 2008. Recruitment took place at Duke and Florida hospitals in the Bone Marrow Transplant clinics during time of clinical appointments in a private location.
Pre-assignment Details: Prior to selecting a donor: donor and subjects had history and physical exam, labs and chest x-ray performed per program and FACT requirements. Female donors should have a negative pregnancy test. Subjects also had bone marrow. Prior to treatment, disease progression and insurance denial led to removal from the study.
Groups:
- Campath Purged Non-myeloablative ASCT: Campath Purged Non-myeloablative allogeneic stem cell transplant (ASCT) in lymphoma, myeloma, or marrow failure: leukemia or myelodysplasia; and solid tumors
  Donor: Will receive granulocyte colony stimulating factor (G-CSF) 10-16 mcg/kg/d subcutaneously(dose will be rounded to the nearest whole vial size and may be divided into bid dosing). Granulocyte-macrophage colony-stimulating factor (GM-CSF) 15 mcg/kg/d subcutaneous or similar growth factor for donor mobilization. Donors will receive at least 3-6 doses of daily growth factor until adequate cells are mobilized.
  Preparative regimen: Begins on day -5 and consist of 4 days of daily fludarabine at 30 mg/m2/d infused over 30 minutes, cyclophosphamide 500 mg/m2/d infused over 1 hour, 5 days of Campath-1H at 20 mg/d in 250 ml of D5 normal saline or normal saline infused over 3 hours.
  Patient Evaluation: Will occur 2-3 times per week by physical exam for toxicity through day 45.
Period: Overall Study
Arm/Group | Campath Purged Non-myeloablative ASCT | Donor Apheresis
Started | 88 | 88
Completed | 78 | 88
Not Completed | 10 | 0
Not completed — Toxicity | 10 | 0

BASELINE CHARACTERISTICS:
Population: Cohort of patients who actually received at least 1 donor lymphocyte infusion (DLI). DLI dosages thus ranged from 1×104 CD3+ cells/kg to 3.27 ×108 CD3+ cells/kg.
Groups:
- Campath Purged Non-myeloablative ASCT: Campath Purged Non-myeloablative ASCT in lymphoma, myeloma, or marrow failure: leukemia or myelodysplasia; and solid tumors
  Donor: Will receive granulocyte colony stimulating factor (G-CSF) 10-16 mcg/kg/d subcutaneously (dose will be rounded to the nearest whole vial size and may be divided into twice daily dosing). Granulocyte macrophage colony stimulating factor (GM-CSF) 15 mcg/kg/d sc or similar growth factor for donor mobilization. Donors will receive at least 3-6 doses of daily growth factor until adequate cells are mobilized.
  Preparative regimen: Begins on day -5 and consist of 4 days of daily fludarabine at 30 mg/m2/d infused over 30 minutes, cyclophosphamide 500 mg/m2/d infused over 1 hour, 5 days of Campath-1H at 20 mg/d in 250 ml of D5 normal saline or normal saline infused over 3 hours.
  Patient Evaluation: Will occur 2-3 times per week by physical exam for toxicity through day 45.
Arm/Group | Campath Purged Non-myeloablative ASCT
Number analyzed (Participants) | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 80
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 54
Region of Enrollment [Number; unit: participants]
  United States | 88

OUTCOME MEASURES:

1. Primary Outcome: Toxicity
Description: Acute graft versus host disease (GVHD) was graded according to the consensus criteria and common terminology criteria (CTC) v3.0 was used for all other toxicities. Recognizing that acute GVHD pathology in the non-ablative and donor lymphocyte infusion (DLI) setting may occur late, we tabulated skin, gut and liver toxicity consistent with acute GVHD (aGVHD) at anytime in the year following the infusion as aGVHD. Toxicities were formally recorded for all patients twice weekly for the first 100 days, at each follow up visit, and as needed intercurrently.
Time Frame: 1 year
Population: Cohort of subjects on the study who received >/=1 donor lymphocyte infusion (DLI). DLI doses thus ranged from 1×104 CD3+ cells/kg to 3.27 ×108 CD3+ cells/kg. Subjects were considered evaluable from the day of first donor lymphocyte (DLI) infusion. Results are not exclusive.
Measure: Number; unit: participants
Groups:
- Campath Purged Non-myeloablative ASCT: Campath Purged Non-myeloablative allogeneic stem cell transplant (ASCT) in lymphoma, myeloma, or marrow failure: leukemia or myelodysplasia; and solid tumors
  Donor: Will receive granulocyte colony stimulating factor (G-CSF) 10-16 mcg/kg/d subcutaneously (dose will be rounded to the nearest whole vial size and may be divided into twice daily dosing). Granulocyte-macrophage colony-stimulating factor (GM-CSF) 15 mcg/kg/d subcutaneous or similar growth factor for donor mobilization. Donors will receive at least 3-6 doses of daily growth factor until adequate cells are mobilized.
  Preparative regimen: Begins on day -5 and consist of 4 days of daily fludarabine at 30 mg/m2/d infused over 30 minutes, cyclophosphamide 500 mg/m2/d infused over 1 hour, 5 days of Campath-1H at 20 mg/d in 250 ml of D5 normal saline or normal saline infused over 3 hours.
  Patient Evaluation: Will occur 2-3 times per week by physical exam for toxicity through day 45.
Arm/Group | Campath Purged Non-myeloablative ASCT
Number analyzed (Participants) | 86
participants
  Acute Graft versus Host Disease (aGvHD) | 5
  Sepsis | 3
  Infection | 10
  Graft Failure | 17
  Cardiac | 3
  Multi-organ failure | 1
  Hepatic Veno-Occlusive Disease | 1
  Post-transplant lymphoproliferative disorder | 2
  Acute respiratory distress syndrome | 2

2. Primary Outcome: Overall Survival (OS)
Description: Estimate toxicity and overall survival rates in subjects treated with a non-myeloablative preparative regimen followed by matched related allogeneic stem cells for allogeneic transplantation.
Time Frame: 8 years
Population: Subjects who completed CAMPATH regimen + 45 days, until disease progression, or death.
Measure: Mean (Full Range); unit: months
Arm/Group | Campath Purged Non-myeloablative ASCT
Number analyzed (Participants) | 78
months | 20 [0.03 to 101]

3. Secondary Outcome: Response
Description: Response Assessment included physical exam and evaluation of peripheral blood and bone marrow. There's no widely accepted criteria for response other than complete response (CR). CR for malignant hematologic diseases is met if all the following are met for >/= 1 month: a) absence of pathologic lymphadenopathy by physical and radiographic exam b) absence of constitutional symptoms due to disease c) Polymorphonuclear leukocyte count >1,500/uL; platelet count >50,000/uL; and hemoglobin >10.0 g/dL d) bone marrow aspirate/biopsy done after (a) through (c) have been met, >/= 30% cellularity and an absence of abnormal lymphoid nodules or cells by flow cytometry, cytogenetics, etc. e) molecular markers of disease must be negative by polymerase chain reaction, Fluorescence in situ hybridization, cytogenetics etc. CR for solid tumors requires complete resolution of disease on physical exam and radiographs. CR for marrow failure is normal white cell, platelet and hematocrit values.
Time Frame: 2 years
Population: Cohort of subjects on the study who actually received >/=1 donor lymphocyte infusion (DLI). DLI doses ranged from 1×104 CD3+ cells/kg to 3.27 ×108 CD3+ cells/kg. Subjects were considered for a second and third DLI 8 weeks apart if they did not have >grade 2 toxicity from the initial DLI, donor availability, and insurance approved the infusion.
Measure: Mean (Full Range); unit: months
Arm/Group | Campath Purged Non-myeloablative ASCT
Number analyzed (Participants) | 88
months
  Partial Response | 4.5 [3 to 6]
  Complete Response | 6 [4 to 19]

ADVERSE EVENTS:
Time Frame: From the beginning of Campath regimen until 6 years after transplant.
Groups:
- Campath Purged Non-myeloablative ASCT: Campath Purged Non-myeloablative ASCT in lymphoma, myeloma, or marrow failure: leukemia or myelodysplasia; and solid tumors
  Donor: Will receive granulocyte colony stimulating factor (G-CSF) 10-16 mcg/kg/d subcutaneously (dose will be rounded to the nearest whole vial size and may be divided into twice daily dosing). Granulocyte macrophage colony stimulating factor (GM-CSF) 15 mcg/kg/d subcutaneously or similar growth factor for donor mobilization. Donors will receive at least 3-6 doses of daily growth factor until adequate cells are mobilized.
  Preparative regimen: Begins on day -5 and consist of 4 days of daily fludarabine at 30 mg/m2/d infused over 30 minutes, cyclophosphamide 500 mg/m2/d infused over 1 hour, 5 days of Campath-1H at 20 mg/d in 250 ml of D5 normal saline or normal saline infused over 3 hours.
  Patient Evaluation: Will occur 2-3 times per week by physical exam for toxicity through day 45.
Arm/Group | Campath Purged Non-myeloablative ASCT
Serious Adverse Events (participants affected / at risk) | 75/88
Other Adverse Events (participants affected / at risk) | 71/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Campath Purged Non-myeloablative ASCT (N=88)
Death (General disorders) | 71 (71)
Hemorrhage (Blood and lymphatic system disorders) | 12 (13)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Campath Purged Non-myeloablative ASCT (N=88)
Failure to Engraft (Blood and lymphatic system disorders) | 16 (17)
Cardiac Left Ventricular Function (Blood and lymphatic system disorders) | 6 (7)
Rash / desquamation (Blood and lymphatic system disorders) | 6 (6)
Diarrhea (Blood and lymphatic system disorders) | 9 (10)
Vomiting (Blood and lymphatic system disorders) | 5 (5)
Febrile Neutropenia (Blood and lymphatic system disorders) | 29 (36)
Infection - other (Infections and infestations) | 10 (10)
Infection - with grade 3 or 4 neutrophils (Infections and infestations) | 35 (65) — Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L)
Infection - grade 1 or 2 neutrophils (Infections and infestations) | 12 (25) — Infection with Grade1 or 2 neutrophils (normal ANC)
Infection - without febrile neutropenia (Infections and infestations) | 30 (64)
Metabolic - Creatinine (Metabolism and nutrition disorders) | 7 (7)
Seizure (Nervous system disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (8) — Shortness of breath
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 14 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No